CLINICAL TRIAL: NCT06390592
Title: Clinical Performance of the Therapy Option FlexPoint (Flexible Volume and Dwell Time Management) of the PD Cycler Sleep•Safe Harmony
Brief Title: Clinical Performance of the Therapy Option FlexPoint of the PD Cycler Sleep•Safe Harmony
Acronym: FlexPoint
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Alcedis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PD-SSH-01-INT
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Renal Failure; Chronic Kidney Disease
Keywords: Renal replacement therapy; Peritoneal dialysis; Automated peritoneal dialysis; PD cycler
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, multi-centric, controlled, randomized, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peritoneal dialysis (PD) (Other): During the clinical phase, patients are treated continuously with the PD cycler sleep•safe harmony.
  The total duration of the clinical phase is six weeks and is divided into 3 Phases à 2 weeks (Clinical phase I, II, and III) which only differ in the FlexPoint settings.
  According to their randomization the patients are treated with Treatment A, B or C in a different order:
  * standard (default) FlexPoint settings (Treatment A)
  * minimum value FlexPoint settings (Treatment B)
  * maximum value for permitted peritoneal residual volume (50%) of FlexPoint settings (Treatment C)
  Interventions: Device: PD cycler

INTERVENTIONS:
Device: PD cycler — Patients are treated continuously during Peritoneal dialysis with the PD cycler sleep•safe harmony with different FlexPoint settings.
  According to their randomization the patients are treated with Treatment A, B or C in a different order:
  * standard (default) FlexPoint settings (Treatment A)
  * minimum value FlexPoint settings (Treatment B)
  * maximum value for permitted peritoneal residual volume (50%) of FlexPoint settings (Treatment C)

SUMMARY:
Analysis and comparison of treatments with and without the FlexPoint technology (flexible volume and dwell time management) of the PD cycler sleep•safe harmony

DETAILED DESCRIPTION:
The primary objective of this study are:

* to investigate and compare the clinical performance of standard (default) FlexPoint settings to minimum FlexPoint settings and to the maximum value for permitted peritoneal residual volume of FlexPoint settings of the PD cycler sleep•safe harmony in the treatment of PD patients.
* to assess whether usage of the settings of the therapy option FlexPoint (flexible volume and dwell time management) of the PD cycler sleep•safe harmony that deviate from the system default and from former sleep•safe settings, influences the efficacy of APD treatments as well as the hydration status (by using BCM) of PD patients.

The secondary objectives of this study are:

* Patients´ Quality of Life (QoL)
* Number of alarms
* To investigate the effects on solute removal
* To investigate the tolerability of the FlexPoint therapy options
* Adverse events / SAE

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by study patient and investigator/ authorised physician
* Minimum age of 18 years
* CKD patients with indication for renal replacement therapy
* Patients being treated with APD for at least 3 months
* Patients using the sleep•safe harmony PD cycler (version 3.1)
* Fluid status regularly monitored with Body Composition Monitor (BCM)
* Proper functioning catheter
* Intraperitoneal Pressure (IPP) ≤ 18 cm H2O
* Ability to understand the nature and requirements of the study

Exclusion Criteria:

* Any conditions which could interference with the patient's ability to comply with the study
* Previous participation in the same study
* Patients who have any condition prohibiting the use of BCM, like patients with major amputations (e.g. lower leg)
* Patients receiving polyglucose containing PD solution
* Respiratory or abdominal wall disease deemed to contraindicate intraperitoneal fill volume (FV) manipulation
* Patients who suffer from peritonitis/exit site infection during the last 4 weeks
* Women of childbearing age without effective means of contraception, pregnancy (pregnancy test will be conducted at start and end of study) or lactation period
* Life expectancy <3 months
* Participation in an interventional clinical study during the preceding 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total Kt/V urea | every 2 weeks, during the 6 weeks treatment
  Measurement of solute removal during peritoneal dialysis focuses on urea

SECONDARY OUTCOMES:
Mean daily ultrafiltration (UF) | every day, during the 6 weeks treatment
  Daily ultrafiltration reached by the patient during peritoneal dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Maite Rivera Gorrín, Dr., Principal Investigator — Hospital Universitario Ramón y Cajal

IPD SHARING:
Plan to Share IPD: No